CLINICAL TRIAL: NCT00491920
Title: High Dosage Vitamin D in the Treatment of Osteoporosis in Postmenopausal Women
Brief Title: High Dosage Vitamin D and Osteoporosis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospital of North Norway (Other)
Collaborators: Norske Kvinners Sanitetsforening Troms (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2006-003186-14
Record Dates: First submitted 2007-06-25; First posted 2007-06-26 (Estimated); Last update posted 2011-11-03 (Estimated); Status verified 2011-11

CONDITIONS: Osteoporosis; Osteopenia
Keywords: osteoporosis; bone mineral density; vitamin D
MeSH Terms: conditions — Osteoporosis; Bone Diseases, Metabolic | interventions — Cholecalciferol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: cholecalciferol (Vitamin D3) — 20 000 Iu x2/week
  + calcium 500 mg/cholecalciferol 400 IU x2/d
Drug: placebo — Calcium 500 mg/Cholecalciferol 400 IU x2/d and placebo 2/w

SUMMARY:
Vitamin D and calcium are essential in the treatment and prevention of osteoporosis. What dosage of vitamin D which is the ideal one, is not yet clear. We want to test the hypothesis that high dosage of vitamin D (i.e. 6500 IU/d) is better than standard dosage (800 IU/d) in a randomized double-blind trial. We will include 400 postmenopausal otherwise healthy women with T-score <= -2.0 in L2-4 or mean total hip. Everybody will receive calcium 1000 mg and vitamin D 800 IU every day. Half of the group will also receive vitamin D 40 000 IU/week, while the other half will have placebo. The study period is one year.

ELIGIBILITY:
Inclusion Criteria:

* bone mineral density in L2-4 or mean total hip with T-score <= -2.0

Exclusion Criteria:

* current use of bisphosphonates, PTH-analogs, estrogen, SERM, p.o. steroids or use of any of these agents last year
* serum creatinin >110 umol/L
* systolic blood pressure >175 mmHg or diastolic blod pressure >105
* serious disease (heart failure, angina pectoris, myocardial infarction, diabetes, mental reduction, granulomatous disease like sarcoidosis, cancer)
* kidney stone
* serum calcium > 2.55 mmol/L
* suspect primary hyperparathyroidism with serum calcium >2.50 mmol/L combined with PTH > 5.0 mmol/L or serum calcium > 2.45 mmol/L combined with PTH >= 7.0 pmol/L

Ages: 50 Years to 80 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 297 (Actual)
Dates: Start 2007-02; Primary Completion 2010-02 (Actual); Study Completion 2010-02 (Actual)

PRIMARY OUTCOMES:
changes in bone mineral density in columna and total hip. | One year

SECONDARY OUTCOMES:
Muscle strength (hand grip strength and knee extension) | One year
balance (tandem test) | One year
body composition (Dexa) | One year
inflammation markers | One year
calcium and vitamin D metabolism | One year
blood lipids | One year
renal function | One year
telomere length | one year
perception of own health | one year
Urinary tract symptoms | one year
effects of polymorphisms in VDR on the other endpoints | one year
side effects | one year

CONTACTS AND LOCATIONS:
Overall Officials: Rolf Jorde, Ph.D, M.D, Principal Investigator — Medical Dpt, University Hospital of Northern Norway
Locations (1):
- Medical Dpt. B, University Hospital of Northern Norway, Tromsø, Norway